CLINICAL TRIAL: NCT05610852
Title: Prospective Single-Center Randomized Study Of Single-Port Transvesical Partial Prostatectomy Versus High Intensity Focused Ultrasound (HIFU)
Brief Title: Single-Port Transvesical Partial Prostatectomy Versus High Intensity Focused Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE10822
Record Dates: First submitted 2022-10-31; First posted 2022-11-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Prostate Adenocarcinoma; Prostate Cancer
Keywords: High Intensity Focused Ultrasound (HIFU); Single-Port Transvesical Partial Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transvesical Single Port Robotic Partial Prostatectomy (Active Comparator): Participants will have a multiparametric prostate MRI and diagnostic prostate biopsy with confirmed localized prostate tumor prior to Prostatectomy. Prostatectomy consists of a single treatment. All participants will have a postoperative visit at 3 days after surgery, followed by phone calls at 1 week, 2 weeks and 4 weeks, followed by office visits at 6 weeks, 3 months, 6 months, 9 months, 1 year, 2 years and 3 years. Participants will be followed indefinitely as per standard of care.
  Interventions: Procedure: Transvesical Single Port Robotic Partial Prostatectomy
- High-intensity focused ultrasound (HIFU) (Active Comparator): Participants will have a multiparametric prostate MRI and diagnostic prostate biopsy with confirmed localized prostate tumor prior to HIFU. HIFU consists of a single treatment. All participants will have a postoperative visit at 3 days after surgery, followed by phone calls at 1 week, 2 weeks and 4 weeks, followed by office visits at 6 weeks, 3 months, 6 months, 9 months, 1 year, 2 years and 3 years. Participants will be followed indefinitely as per standard of care.
  Interventions: Procedure: High-intensity focused ultrasound (HIFU)

INTERVENTIONS:
Procedure: Transvesical Single Port Robotic Partial Prostatectomy — A foley catheter is inserted on the sterile field. A suprapubic midline incision is made and the da Vinci SP surgical system is docked percutaneously directly to the bladder. Prior to the operation, a radiologist identifies and segments tumors and the urethra. A transrectal ultrasound probe is inserted and secured into a fixed position. The Koelis software is utilized to fuse MRI and ultrasound images to identify the target lesion in real-time, allowing for intraoperative guidance. The ultrasound probe rotates automatically, allowing for localization of the tumor intraoperatively. Then depending on the area of the tumor, a Hemi or quadrant resection is completed while preserving the nerves, vas deferens, and seminal vesicles. The urethrovesical anastomosis is then performed.
  Arms: Transvesical Single Port Robotic Partial Prostatectomy
Procedure: High-intensity focused ultrasound (HIFU) — Three contoured measurements are required for the MR fusion system to reproduce the volume of the prostate. Following this, the area to be targeted will be selected in graded fashion from the anterior to posterior of the prostate. Once planning of ROI (region of interest) is complete, the HIFU treatment may begin. Quadrant or hemi ablation will be performed based on the size and complexity of the tumor. The distal margin of the ablation will be kept at least 4 mm away from the external sphincter. The rectal temperature and its distance from the probe will be carefully monitored throughout the procedure.
  Arms: High-intensity focused ultrasound (HIFU)

SUMMARY:
This study aims to compare the novel single-port robotic partial prostatectomy to High-intensity focused ultrasound (HIFU) in patients with low to intermediate risk localized prostate cancer. These interventions have become acceptable focal therapies prevalent with beneficial oncologic outcomes and therefore need to be examined further.

DETAILED DESCRIPTION:
The primary objective is to evaluate the in-field recurrence rates and recurrence free survival - defined as the absence of clinically significant prostate cancer within the treated zone (identified by prostate MRI and subsequent targeted prostate biopsy).

Secondary objectives of interest are:

* Perioperative parameters such as operative time, perioperative complications, analgesic requirement, postoperative hospital stay, foley catheter duration
* Functional outcomes such as time to urinary continence, urinary continence, and erectile dysfunction
* Oncologic outcomes such as biochemical recurrence rates (defined in section 2.1), recurrence free survival, presence of secondary intervention for prostate cancer (HIFU, radiation, surgery, ADT)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically: Biopsy-confirmed prostate cancer, stage T1a, T2a, T2b, or T2c prostate cancer using MRI staging, with a region of interest (ROI) PIRADs grade 3 or greater, Serum PSA 10 ng/ml or less, Region of interest on MRI of grade 3 or greater
* The MRI performed must include at least:
* A T2-weighted sequence in sections ≤ 4 mm, centered on the prostate and seminal vesicles, at least in the axial plane. Alternatively, a 3D T2-weighted sequence can be realized,
* A diffusion sequence of ≤ 4 mm slice in the axial plane. An ADC card will be provided and calculated from at least two values of b, the maximum value of b being ≥ 600 s / mm2,
* A dynamic sequence after gadolinium injection. It will be a sequence of echo T1-weighted gradient of slice ≤ 4 mm, centered on the prostate and seminal vesicles in the axial plane, with or without fat saturation. A first series will be performed without contrast injection, and will be repeated iteratively for the arrival of a bolus of gadolinium chelates. The time resolution (that is to say, the acquisition time of one dynamic series will be ≤ 20 seconds). The number of chained dynamic series is calculated so that the total length of the dynamic acquisition be at least 3 minutes
* A total dose of 0.1 mmol / kg of gadolinium chelate will be injected at a rate of 3-4 mL / s by using an automatic injector, in a vein of the hand of the forearm or elbow.
* If necessary, subtracted images are calculated
* Clinically significant prostate cancer defined as Gleason score 3+4 or less in any core
* Biopsies for preoperative diagnosis of prostate cancer will have included: At least 12 randomized samples (2 samples per sextant), At least two targeted sampling on each target score MRI ESUR ≥ 3/5
* Life expectancy greater than 10 years.
* Age >18 years.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with any prior extensive pelvic surgery, pelvic fractures, hemorrhoid, fissure surgery, cardiac pacemaker, or metal prosthesis
* Prior treatment for prostate cancer such as radiotherapy, focal or hormonal therapy
* Uncorrected coagulopathy or history of Latex allergy
* Active soft tissue or urinary infection, indwelling Foley catheter or severe irritative or obstructive symptoms
* Poor surgical risk (defined as American Society of Anesthesiology score > 3).
* Any condition or history of illness or surgery that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient (e.g. significant cardiovascular conditions that significantly affect the life expectancy, chronic opiate use, pain syndrome, or drug abuse.)
* Prostate size larger than 80 grams.
* Subjects with prostatic Calcification (>0.5 cc) close to the area to be treated.
* Subjects with extraprostatic extension or cribriform pattern on biopsy.
* Subjectes with sexual dysfunction defined as SHIM score < 17
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival Recurrence free survival | 1 year after treatment
  Number of patients with absence of clinically significant prostate cancer on prostate MRI and targeted prostate biopsy
Recurrence free survival | 2 years after treatment
  Number of patients with absence of clinically significant prostate cancer on prostate MRI and targeted prostate biopsy
Recurrence free survival | 3 years after treatment
  Number of patients with absence of clinically significant prostate cancer on prostate MRI and targeted prostate biopsy

SECONDARY OUTCOMES:
Operative time | At initial treatment (postoperative day 0)
  Minutes from incision to closing during surgery (median)
Postoperative Complications | Within 3 months after treatment.
  Clavien-dindo classification number (1-5), number (percent)
Analgesic requirment | Once at first follow up (up to 7 days after initial treatment)
  Units of oral morphine equivalent dosing (mg), median
Postoperative hospital stay | Up to 1 day after initial treatment
  Time that patient is observed in the hospital after surgery, in hours (median)
Foley catheter duration | Up to 7 days after initial treatment
  Time at which the foley catheter is removed after treatment, in days (median)
Time to urinary continence | Assessed at each visit for up to 1 year after treatment
  Time at which the patient becomes continent in days (median)
Urinary continence | Assessed at each visit for up to 1 year after treatment
  Continence defined as using 1 pad for security or less for stress urinary incontince, recorded as yes or no (percent)
Erectile dysfunction | Assessed at each visit for up to 3 years
  Assessed using scores from a validated survey (IIEF-5). Recorded as the the score from 5 (impotent) to 25 (no impotence), median.
Biochemical recurrence | Assessed at each visit for up to 3 years
  PSA recurrence defined as PSA nadir after treatment +1ng/ml within 12 months or PSA Nadir + 1.5ng/ml from 12-36 months. Recorded as yes or no (percent)
Secondary interventions | Assessed at the time of clinic visits up to 3 years after treatment.
  Time point at which the patient undergoes treatment for prostate cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Kaouk, MD, Principal Investigator — Glickman Urological & Kidney Institute: Professor of Urology
Locations (1):
- Glickman Urological & Kidney Institute, Cleveland Clinic Foundation, Case Comprehensive Cancer Center, Cleveland, Ohio, United States